CLINICAL TRIAL: NCT03820466
Title: Investigator-initiated, Placebo-controlled, Randomized Trial to Assess the Efficacy and Safety of Platelet Inhibition and/ or Lipid Lowering in Non-ACS-patients With Elevated High-sensitivity Troponin Values
Brief Title: Effect of Platelet Inhibition and / or Lipid Lowering in Non-ACS-patients With Positive Troponin
Acronym: GRAY-ZONE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient recruitment due to the pandemic situation
Sponsor: Dr. med. Mahir Karakas (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Mahir Karakas, Coordinating Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GRAY-ZONE
Record Dates: First submitted 2017-10-02; First posted 2019-01-29 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Acute Chest Syndrome
Keywords: Aspirin; Atorvastatin; Troponin
MeSH Terms: conditions — Acute Chest Syndrome | interventions — Aspirin; Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aspirin (Active Comparator): Aspirin 100 mg once daily and Placebo Atorvastatin once daily
  Interventions: Drug: Aspirin; Drug: Placebo Atorvastatin
- Atorvastatin (Active Comparator): Atorvastatin 20 mg once daily and Placebo Aspirin once daily
  Interventions: Drug: Atorvastatin; Drug: Placebo Aspirin
- Aspirin-Atorvastatin (Experimental): Aspirin 100 mg once daily and Atorvastatin 20 mg once daily
  Interventions: Drug: Aspirin; Drug: Atorvastatin
- Placebo (Placebo Comparator): Placebo Aspirin once daily and Placebo Atorvastatin once daily
  Interventions: Drug: Placebo Aspirin; Drug: Placebo Atorvastatin

INTERVENTIONS:
Drug: Aspirin — Once daily application of platelet inhibiting medication
  Other Names: Acetyl Salicyl Acid
  Arms: Aspirin; Aspirin-Atorvastatin
Drug: Atorvastatin — Once daily application of lipid lowering medication
  Other Names: Statin
  Arms: Aspirin-Atorvastatin; Atorvastatin
Drug: Placebo Aspirin — Once daily application of placebo
  Other Names: Placebo Oral Tablet
  Arms: Atorvastatin; Placebo
Drug: Placebo Atorvastatin — Once daily application of placebo
  Other Names: Placebo Oral Tablet
  Arms: Aspirin; Placebo

SUMMARY:
The study evaluates the effect of platelet inhibition and / or lipid lowering in non-ACS-patients with symptoms suggestive for ACS, and elevated high-sensitivity troponin values

DETAILED DESCRIPTION:
Current databases show, that high-/ ultra sensitive (hs)/ (us) troponin levels above the 99th percentile in patients presenting with chest pain are indicative for future cardiovascular events, even when acute coronary syndrome (ACS) was ruled out. Most of these non-ACS-patients are discharged without specific/ preventive therapy (anti-platelet or anti-lipid), although "positive" troponin values (any value at any time during hospitalisation above the 99th percentile) seem to clearly indicate underlying myocardial ischemia. In summary, there is an unmet need and huge potential to reduce mortality and morbidity in Chest Pain Unit patients by specific therapy. The investigators propose that platelet inhibition by Aspirin or lipid lowering by Atorvastatin will prevent plaque rupture and superimposition of thrombosis to coronary atherosclerosis in this population. It is planned to conduct a controlled clinical trial: 3,000 troponin positive patients presenting at emergency room (ER)/ CPU with symptoms suggestive for ACS, but an ACS was ruled out, will be assigned randomly to Aspirin 100 mg and/ or Atorvastatin 20 mg versus placebo (2x2 factorial design).

ELIGIBILITY:
Inclusion Criteria:

* Patient with symptoms suggestive for ACS presenting within 48 hours after onset in the ER/ Chest Pain Unit (CPU)
* Patient has at least one elevated high-sensitivity troponin I or T value
* Chest pain is classified as non-ACS, despite elevated hsTn (e.g. because of missing troponin dynamics)
* At least 50 years of age

Exclusion Criteria:

* Indication for antiplatelet therapy (e.g transient ischemic attack, or stable coronary artery diseases -CAD) or anticoagulation therapy (such as atrial fibrillation)
* Indication for anti-lipid therapy
* Any evidence of an acute myocardial necrosis (e.g imaging evidence of new regional wall motion abnormality, or significant ST-segment-T wave (ST-T) changes in ECG)
* Untreated clinically significant CAD requiring revascularization
* Hemoglobin value below 8 mg/d, and/or creatinine kinase ≥3 times ULN, and/or AST or ALT ≥3 times ULN
* Active malignancy of any organ system, treated or untreated. Subjects have to be in remission for at least 36 months to be eligible.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Myocardial infarction and/ or cardiovascular death and/ or revascularization | Until last patient has completed 12 months of follow-up
  Time to myocardial infarction, coronary revascularization, or death, whatever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Mahir Karakas, MD, Study Chair — University Heart Center Hamburg
Locations (7):
- Germany (7):
  - University of Berlin, Campus Benjamin-Franklin, Berlin
  - Asklepios Harz-Hospital Goslar, Goslar
  - University Heart Center Hamburg, Hamburg
  - University of Heidelberg, Heidelberg
  - University of Leipzig, Leipzig
  - Robert-Bosch-Hospital Stuttgart, Stuttgart
  - University of Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No